CLINICAL TRIAL: NCT03493321
Title: Role of PRF With MTA and Theracal After Pulpotomy in Relieving Pain and Maintaining the Vitality of the Remaining Radicular Pulp Tissue in Permanent Posterior Teeth With Closed Root Apices: "Randomized Controlled Trial"
Brief Title: Role of PRF With MTA and Theracal After Pulpotomy in Relieving Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Essam, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-03-07
Record Dates: First submitted 2018-03-12; First posted 2018-04-10 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Neuritis
MeSH Terms: conditions — Neuritis | interventions — Prolactin-Releasing Hormone; TheraCal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRF with MTA (Experimental): PRF with MTA with PRF with Theracal as intervention
  Interventions: Other: PRF with Theracal

INTERVENTIONS:
Other: PRF with Theracal — using the PRF which is a new technique with an bioactive material which is the Theracal to evaluate its effect upon the radicular pulp tissue

SUMMARY:
this research will evaluate the effect of PRF with different bioactive materials in dentistry

DETAILED DESCRIPTION:
PRF will be used with MTA and Theracal to evaluate its effect upon these materials in reliving pain and maintains the teeth vitality in permanent teeth with closed apices, in order to improve the materials outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Symptomatic pulpitis.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow-up period.
* Patients with mature root.
* Patients with no periapical lesion.
* Patients with localized pain.
* Posterior teeth only will be involved

Exclusion Criteria:

* Patients with immature roots.
* Patients with any systemic disease that may affect normal healing.
* Patients with periapical lesions or infections.
* Pregnant females.
* Patients who could/would not participate in a 1-year follow-up.
* Patients with fistula.
* Patients with necrotic pulp.
* Patients with old age.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-08-22 (Estimated); Primary Completion 2019-08-22 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
pain after the process | 1 year
  Questionnaire by asking the patient about the pain intensity

SECONDARY OUTCOMES:
dentin bridge formation | 1 year
  X-ray
no periapical radiolucency | 1 year
  X-ray